CLINICAL TRIAL: NCT03365401
Title: Surgical Treatment Versus Nonoperative Treatment in Lumbar Spinal Stenosis: a Multicenter Open-label Randomized Controlled Trial
Brief Title: Efficiency of Surgical Treatment for Lumbar Spinal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Liu Haiying, department of spinal surgery, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSS011
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Lumbar Spinal Stenosis
Keywords: surgery; decompression
MeSH Terms: conditions — Spinal Stenosis | interventions — Laminectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grade 1 (Experimental): Decompression surgery
  Interventions: Procedure: decompression surgery
- grade 2 (Active Comparator): nonsurgical treatment
  Interventions: Procedure: nonsurgical treatment

INTERVENTIONS:
Procedure: decompression surgery — undertake decompression surgery
  Arms: grade 1
Procedure: nonsurgical treatment — complete on bed with prevention of complication
  Arms: grade 2

SUMMARY:
Decompression surgery has proved to be effective for Lumbar Spinal Stenosis (LSS) with persistent pain. But the efficiency of the surgery for degenerated LSS remain uncertain and is the subject of this study. This is a multiple center open-label randomised trial. Patients were randomly allocated to surgical group or a nonoperative group. Because of the procedure , neither patients nor investigators were blinded. The primary outcome is the change of symptom measure by the Oswestry disability index 6, 12, and 24 months after procedure.

DETAILED DESCRIPTION:
This study will use a randomised controlled trial to access the efficiency of the surgery for degenerated LSS. Patients aged 50 years or older, had LSS will be invited to take part. Patients will be randomised divided into 2 arms. The participants in the intervention arm will have decompression surgery ; those randomised to the control arm will receive current standard conservative treatment methods.

Patients were clinically assessed at baseline (the day of surgery or treatment), and at 6,12 and 24 months afterwards. The primary outcome will be the pain release , categorised according to Oswestry disability index.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptoms: back pain radiation to lower limbs or buttocks; fatigue or loss of sensation in the lower limbs aggravated by walking.
* Persistent pain without progressive neurologic dysfunction
* Duration of symptoms and signs for more than 6 months
* Severity of the disease justifying either surgical or nonoperative treatment

Exclusion Criteria:

* severe LSS with intractable pain and progressive neurologic dysfunction, suggesting forthcoming surgical treatment
* spinal stenosis not caused by degeneration
* lumbar herniated disc diagnosed during the last 12 months
* neurologic disease causing impaired function of the lower limbs

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-02-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
change of symptoms | 6, 12, and 24 months
  Oswestry disability index (ODI)

SECONDARY OUTCOMES:
change of pain relief | 6, 12, and 24 months
  World Health Organization pain classification

CONTACTS AND LOCATIONS:
Overall Officials: haiying liu, Study Director — pekingUPH department of spinal surgery

IPD SHARING:
Plan to Share IPD: No